CLINICAL TRIAL: NCT06607627
Title: An Open-Label, Single-arm Study to Evaluate the Pharmacokinetics (PK), Pharmacodynamics (PD), Safety, and Efficacy of Gefurulimab in Pediatric Patients (6 to < 18 Years of Age) With Generalized Myasthenia Gravis (gMG) Who Express Acetylcholine Receptor Antibodies (AChR+)
Brief Title: PK, PD, Safety, and Efficacy Study of Gefurulimab in Pediatric Patients With AChR+ Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6780C00004; 2024-515157-17-00 (Other: EUCT); ALXN1720-MG-302 (Other: Alexion); U1111-1327-6615 (Other: WHO)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Generalized Myasthenia Gravis; gMG
Keywords: Acetylcholine Receptor antibodies; AChR+; Generalized Myasthenia Gravis; gMG; ALXN1720; anti-acetylcholine receptor antibody-positive; acetylcholine receptor; AChR; myasthenia gravis; MG; complement component 5; C5; VHH antibody; pediatric
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Gefurulimab (Experimental): On Day 1, participants will receive a weight based loading dose followed by a weekly maintenance dose for up to 122 weeks.
  Interventions: Combination Product: Gefurulimab

INTERVENTIONS:
Combination Product: Gefurulimab — Combination product consisting of syringe prefilled with gefurulimab will be administered weekly via subcutaneous (SC) injection.

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics and pharmacodynamics of gefurulimab in pediatric participants with AChR+ gMG for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

United States of America (USA) specific inclusion criterion:

* Participant must be 12 to < 18 years of age at the time of signing the informed consent/assent.
* All participants must be vaccinated against meningococcal infection from serogroups A, B, C, W, and Y within 3 years and at least 2 weeks prior to the first dose of study intervention administration.

Rest of World (ROW) specific inclusion criteria:

* Participant must be 6 to < 18 years of age at the time of signing the informed consent/assent.
* All participants must be vaccinated against meningococcal infection from serogroups A, C, W, Y (and B where available) within 3 years prior to study intervention on Day 1. If vaccination occurs < 2 weeks prior to Day 1, the participants will receive prophylactic antibiotics for at least 2 weeks after initial meningococcal vaccination for serogroups A,C,W,Y (and B, where available)

Global inclusion criteria:

* Diagnosis of MG with generalized muscle weakness meeting the clinical criteria defined by Myasthenia Gravis Foundation of America (MGFA) Class II, III or IV
* Positive serological test for autoantibodies against AChR

Exclusion Criteria:

* History of thymectomy, or any other thymic surgery within 12 months prior to Screening
* Untreated thymic malignancy, carcinoma, or thymoma
* History of Neisseria meningitidis infection
* Pregnancy, breastfeeding, or intention to conceive during the course of the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2029-01-23 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Gefurulimab | Day 1 predose through Week 18 predose
Serum Free Complement Component 5 (C5) Concentration | Day 1 predose through Week 18 predose

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day 1 through Week 134
Change in Quantitative Myasthenia Gravis Score for Disease Severity (QMG) Total Score From Baseline Through Week 18 | Baseline through Week 18
Number of Participants With ≥ 5-point Reduction From Baseline in the QMG Total Score Through Week 18 | Baseline through Week 18
Change in Myasthenia Gravis Activities of Daily Living Profile (MG-ADL) Total Score From Baseline Through Week 18 | Baseline through Week 18
Number of Participants With ≥ 3-point Reduction From Baseline in the MG-ADL Total Score Through Week 18 | Baseline through Week 18
Number of Participants With Anti-drug Antibodies (ADAs) | Baseline through Week 134
Number of ADA Positive Participants With Pre-existing Immunoreactivity,Treatment-emergent or Treatment-boosted ADA Responses | Baseline through Week 134
Number of ADA Positive Participants With Neutralizing Antibody (NAb) Positive or Negative Status | Baseline through Week 134

CONTACTS AND LOCATIONS:
Locations (12):
- United States (2):
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Norfolk, Virginia
- Brazil (4):
  - Research Site, Joinville
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Research Site, Saitama-shi, Japan
- Poland (3):
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Warsaw
- Taiwan (2):
  - Research Site, New Taipei City
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR